CLINICAL TRIAL: NCT01061697
Title: Open Labelled Study of Pregabalin in the Treatment of Neuropathic Pain in Cervical Myeloradiculopathy (Pregabalin and Radicular Pain Study (PARPS))
Brief Title: Pregabalin and Radicular Pain Study (PARPS)
Acronym: PARPS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: A/Prof Lo Yew Long, National Neuroscience Institute, Singapore General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #2006/072/A
Record Dates: First submitted 2010-02-02; First posted 2010-02-03 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2011-07

CONDITIONS: Cervical Spondylosis; Cervical Spondylotic Myelopathy; Cervical Spondylotic Radiculopathy
MeSH Terms: conditions — Spondylosis | interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Pregabalin — At week 0, pregabalin 75mgbd will be given for 1 month. If visual analogue scale is not reduced by 50% after 1 month, pregabalin will be increased to 150mgbd for the second month
  Other Names: Brand name: Lyrica

SUMMARY:
This study is designed to investigate the effectiveness of pregabalin (Lyrica) on nerve pain caused by degenerative neck problems. Pregabalin is a new drug registered for use in nerve pain worldwide

DETAILED DESCRIPTION:
The treatment of neuropathic pain is clinically challenging, and pain from cervical spondylosis (CS) is a common variant. This may result from degenerative spinal canal/cord stenosis (cervical spondylotic myelopathy (CSM)) or lateral recesses compromise, leading to nerve root compression (cervical spondylotic radiculopathy (CSR)).

Pregabalin is a newly registered drug for the treatment of neuropathic pain. Its efficacy has been proven in randomised, placebo-controlled trials for post-herpetic neuralgia and diabetic neuropathy. However, its efficacy in CS with underlying CSR or CSM has not been established. Additionally, there are no data to date on its use in Asian patients.

In this study, we prospectively evaluate its efficacy for treating neuropathic pain in degenerative CSR/ CSM 60 patients in an open-labelled, add on fashion. Self-evaluation and investigator rated scoring will be implemented.

The results will be of value in the non-operative management of CS.

ELIGIBILITY:
Inclusion Criteria:

* Clinical & MRI, or electrophysiological evidence of pain due to radiculopathy
* Patients with CS and CSR or CSM with neuropathic pain due to the above in the neck and upper limbs or lower limbs (including dysesthesia, paresthesia, hyperalgesia).

Exclusion Criteria:

* Diabetic neuropathy or other underlying neuropathic conditions
* Contraindications and allergy to pregabalin
* Previously treated with gabapentin in the last 8 weeks
* Pregnant or breast feeding
* History of renal impairment
* History of other causes of neuropathic pain

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-01; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS): Pain ruler done daily | 2 months

SECONDARY OUTCOMES:
Short-Form McGill Pain Questionnaire (SFMPQ) | 0, 1, 2 months
Patient and Clinical Global Impression of change | 0, 1, 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Y L Lo, MD, Principal Investigator — National Neuroscience Institute, Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Outram Road, Singapore